CLINICAL TRIAL: NCT04498611
Title: Prediction of Upgrade to Invasive Cancer in Patients Diagnosed With Ductal Carcinoma in Situ by Percutaneous Core Needle Biopsy: A Development and Validation Study
Brief Title: Prediction of Upgrade to Invasive Cancer in Patients Diagnosed With Ductal Carcinoma in Situ by Percutaneous Core Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-219-1119
Record Dates: First submitted 2020-07-14; First posted 2020-08-04 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Ductal, Breast; Invasive Breast Cancer; IMAGE
MeSH Terms: conditions — Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breast DCIS patients (Experimental): Breast DCIS patients who diagnosed by tissue biopsy except excisional biopsy before surgery, and who agreed to taking the breast MRI.
  Interventions: Diagnostic Test: contrast-enhanced breast MRI

INTERVENTIONS:
Diagnostic Test: contrast-enhanced breast MRI — Contrast-enhanced MRI will be performed on patients diagnosed with ductal carcinoma in-situ (DCIS) by preoperative biopsy.

SUMMARY:
It is considered that whether or not the accompanying invasive cancer classified through MRI images of breast cancer patients identified as Ductal Carcinoma in situ (DCIS) through preoperative tissue biopsy is significantly consistent with the postoperative stage.

Therefore, this study intend to evaluate the effectiveness as a diagnostic tool that can help determine the axillary lymph node surgery by predicting the possibility of post-operative up-staging using magnetic resonance imagings of breast cancer patients who have been identified as ductal carcinoma in situ and are scheduled for surgery.

DETAILED DESCRIPTION:
1. To date, there is no significant research data on the value of the Apparent Diffusion Coefficient (ADC) that can distinguish between pure Ductal Carcinoma in situ (pure DCIS) and invasive cancer (DCIS-IC), from June 2019 to 2020 1 Of the 144 patients who obtained Diffusion Weighted images (b=0,800,1200) with 3.0-T MRI equipment and diagnosed with ductal carcinoma in situ on the biopsy, among 144 patients who did not undergo preoperative chemotherapy using a CAD program, the 3-dimensional Apparent Diffusion Coefficient value of the tumor is measured and compared with whether or not there is invasive cancer after surgery, and the optimal Apparent Diffusion Coefficient reference value that can predict the invasive cancer will be retrospectively derived.
2. Scheduled MRI tests will be performed on patients enrolled from July 2020, and will be performed using the standard protocols (3T, contrast enhancement and diffuse enhancement images DWI b0,800,1200). Among the MRI images taken, the range of lesions is evaluated in contrast-enhanced T1-highlighted images, and the Apparent Diffusion Coefficient values of the lesions are three-dimensionally mapped using a CAD program and histogram analysis on diffused images. The ADC reference value derived from the retrospective analysis is used to predict prospectively for invasive cancer in all lesions.
3. Mastectomy is performed according to the existing surgical method. Axillary lymph node surgery is determined according to the existing decision method (tumor location, size, range, histological grade, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Adult over 19 years-old
* Breast Ductal Carcinoma in-situ patients who diagnosed preoperative tissue biopsy
* A person who understands this study and agrees with willingness to participate

Exclusion Criteria:

* Ductal Carcinoma in-situ which diagnosed excisional biopsy
* When there is no lesion that can be discriminated from magnetic resonance imaging
* Neoadjuvant chemotherapy patients
* Patients who have complication (hematoma, abscess etc.) after preoperative biopsy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Comparing of Preoperative MRI and Postoperative histopathologic results | 2 weeks after surgery
  Analysis of the concordance rate (%) of invasive cancers confirmed in the final histopathology after surgery.

SECONDARY OUTCOMES:
Comparing the predicted upstaging rate through the MRI and histopathologic results | 3 weeks after surgery
  Analysis the proportion of up-staging(%) of invasion cancer in the final histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Gon Moon, Study Director — Seoul National University of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- [Background] Mori N, Ota H, Mugikura S, Takasawa C, Tominaga J, Ishida T, Watanabe M, Takase K, Takahashi S. Detection of invasive components in cases of breast ductal carcinoma in situ on biopsy by using apparent diffusion coefficient MR parameters. Eur Radiol. 2013 Oct;23(10):2705-12. doi: 10.1007/s00330-013-2902-2. Epub 2013 Jun 4. PMID 23732688
- [Background] Baxter GC, Graves MJ, Gilbert FJ, Patterson AJ. A Meta-analysis of the Diagnostic Performance of Diffusion MRI for Breast Lesion Characterization. Radiology. 2019 Jun;291(3):632-641. doi: 10.1148/radiol.2019182510. Epub 2019 Apr 23. PMID 31012817
- [Background] Surov A, Meyer HJ, Wienke A. Can apparent diffusion coefficient (ADC) distinguish breast cancer from benign breast findings? A meta-analysis based on 13 847 lesions. BMC Cancer. 2019 Oct 15;19(1):955. doi: 10.1186/s12885-019-6201-4. PMID 31615463
- [Background] Lamb LR, Lehman CD, Oseni TO, Bahl M. Ductal Carcinoma In Situ (DCIS) at Breast MRI: Predictors of Upgrade to Invasive Carcinoma. Acad Radiol. 2020 Oct;27(10):1394-1399. doi: 10.1016/j.acra.2019.09.025. Epub 2019 Nov 4. PMID 31699638
- [Background] Lee KH, Han JW, Kim EY, Yun JS, Park YL, Park CH. Predictive factors for the presence of invasive components in patients diagnosed with ductal carcinoma in situ based on preoperative biopsy. BMC Cancer. 2019 Dec 10;19(1):1201. doi: 10.1186/s12885-019-6417-3. PMID 31822268
- [Background] Borlinhas F, Conceicao RC, Ferreira HA. Optimal b-values for diffusion kurtosis imaging in invasive ductal carcinoma versus ductal carcinoma in situ breast lesions. Australas Phys Eng Sci Med. 2019 Sep;42(3):871-885. doi: 10.1007/s13246-019-00773-2. Epub 2019 Jul 18. PMID 31321627